CLINICAL TRIAL: NCT03085095
Title: HERO: A Multinational Phase 3 Randomized, Open-label, Parallel Group Study to Evaluate the Safety and Efficacy of Relugolix in Men With Advanced Prostate Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Relugolix in Men With Advanced Prostate Cancer
Acronym: HERO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-3201; 2017-000160-15 (EudraCT Number)
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relugolix (Experimental): Relugolix for 48 weeks
  Interventions: Drug: Relugolix
- Leuprolide Acetate (Active Comparator): Leuprolide acetate for 48 weeks
  Interventions: Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Relugolix — Relugolix 120-mg tablet administered orally once daily following an oral loading dose of 360 mg (3 x 120-mg tablets) on Day 1
  Other Names: TAK-385; MVT-601; RVT-601; T-1331285
  Arms: Relugolix
Drug: Leuprolide Acetate — Leuprolide acetate depot suspension, 22.5 mg (or 11.25 mg in Japan, Taiwan, and China), every 3 months by subcutaneous injection
  Other Names: Leuprolide
  Arms: Leuprolide Acetate

SUMMARY:
The purpose of this study is to determine the efficacy and safety of relugolix 120 milligrams (mg) orally once daily for 48 weeks on maintaining serum testosterone suppression to castrate levels (< 50 nanograms/deciliter [ng/dL]) in participants with androgen-sensitive advanced prostate cancer.

DETAILED DESCRIPTION:
This is a phase 3, multinational, randomized, open-label, parallel group study to evaluate the efficacy and safety of oral daily relugolix 120 mg in participants with androgen-sensitive advanced prostate cancer who require at least 1 year of continuous androgen-deprivation therapy. Relugolix 120 mg orally once daily or leuprolide acetate depot suspension, 22.5 mg (or 11.25 mg in Japan and Taiwan based on local labels), every 3 months by subcutaneous injection will be administered to participants.

There are 2 analyses for this study, a primary analysis and a final analysis.

Primary Analysis:

The primary analysis of efficacy and safety has been completed (N=934). Participants were randomized 2:1 to receive relugolix or leuprolide for 48 weeks, followed by a 30-day safety follow-up visit or early termination 30-day safety follow-up.

Final Analysis:

The final analysis will occur after additional participants with metastatic disease (approximately 130) have been enrolled and randomized from any sites to the study, and have completed the 48-week treatment period. A cohort of participants enrolled in China and Taiwan will be analyzed separately once they have completed treatment to support registration in China.

Eligible participants were randomized 2:1 to relugolix or leuprolide arm and will attend visits monthly (every 4 weeks) where serum testosterone and prostate-specific antigen will be assessed. Safety will be assessed throughout the study by monitoring adverse events, vital signs, physical examinations, clinical laboratory tests, and 12-lead electrocardiograms.

Castration resistance-free survival will be assessed up to Week 49, Day 1 of the study and reported as part of the final analysis.

The study enrolled 1134 participants, including 139 participants with metastatic advanced prostate cancer to support the analysis of the secondary endpoint of castration resistance-free survival and 93 Chinese participants (enrolled in China and Taiwan) to support registration in China.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate.
2. Is a candidate for, in the opinion of the investigator, at least 1 year of continuous androgen deprivation therapy for the management of androgen-sensitive advanced prostate cancer with 1 of the following clinical disease state presentations:

   1. Evidence of biochemical (PSA) or clinical relapse following local primary intervention with curative intent, such as surgery, radiation therapy, cryotherapy, or high-frequency ultrasound and not a candidate for salvage treatment by surgery; or
   2. Newly diagnosed androgen-sensitive metastatic disease; or
   3. Advanced localized disease unlikely to be cured by local primary intervention with either surgery or radiation with curative intent.
3. Has a serum testosterone at the Screening visit of ≥ 150 ng/dL (5.2 nanomoles [nmol]/liter [L]).
4. Has a serum PSA concentration at the Screening visit of > 2.0 ng/milliliter (mL) (2.0 microgram [μg]/L), or, when applicable, post radical prostatectomy of > 0.2 ng/mL (0.2 μg/L) or post radiotherapy, cryotherapy, or high frequency ultrasound > 2.0 ng/mL (2.0 μg/L) above the post interventional nadir.
5. Has an Eastern Cooperative Oncology Group performance status of 0 or 1 at initial screening and at baseline.

Key Exclusion Criteria:

1. In the investigator's opinion, is likely to require chemotherapy or surgical therapy for symptomatic disease management within 2 months of initiating androgen deprivation therapy.
2. Previously received gonadotropin-releasing hormone analog or other form of androgen deprivation therapy (estrogen or antiandrogen) for > 18 months total duration. If androgen deprivation therapy was received for ≤ 18 months total duration, then that therapy must have been completed at least 3 months prior to baseline. If the dosing interval of the depot is longer than 3 months, then the prior androgen deprivation therapy must have been completed at least as long as the dosing interval of the depot.
3. Previous systemic cytotoxic treatment for prostate cancer (for example, taxane-based regimen).
4. Metastases to brain per prior clinical evaluation.
5. Participants with myocardial infarction, unstable symptomatic ischemic heart disease, cerebrovascular events, or any significant cardiac condition within the prior 6 months.
6. Active conduction system abnormalities.
7. Uncontrolled hypertension.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2021-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Monitor, Study Director — Myovant Sciences
Locations (151):
- United States (27):
  - Tucson, Tucson, Arizona
  - Orange, Orange, California
  - Denver, Denver, Colorado
  - Pompano Beach, Pompano Beach, Florida
  - Jeffersonville, Jeffersonville, Indiana
  - Des Moines, Des Moines, Iowa
  - Wichita, Wichita, Kansas
  - Baltimore, Baltimore, Maryland
  - Troy, Troy, Michigan
  - Omaha, Omaha, Nebraska
  - Las Vegas, Las Vegas, Nevada
  - Brick, Brick, New Jersey
  - Albuquerque, Albuquerque, New Mexico
  - Albany, Albany, New York
  - Garden City, Garden City, New York
  - Plainview, Plainview, New York
  - Poughkeepsie, Poughkeepsie, New York
  - Syracuse, Syracuse, New York
  - Durham, Durham, North Carolina
  - Greensboro, Greensboro, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Middleburg Heights, Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma City, Oklahoma
  - Lancaster, Lancaster, Pennsylvania
  - Myrtle Beach, Myrtle Beach, South Carolina
  - Nashville, Nashville, Tennessee
  - San Antonio, San Antonio, Texas
- Australia (5):
  - Camperdown, Camperdown, New South Wales
  - Tweed Heads, Tweed Heads, New South Wales
  - Wahroonga, Wahroonga, New South Wales
  - Redcliffe, Redcliffe, Queensland
  - Southport, Southport, Queensland
- Linz, Linz, Austria
- Belgium (3):
  - Gent, Ghent, Oost-Vlaanderen
  - Brussels, Brussels
  - Kortrijk, Kortrijk
- Brazil (10):
  - Itabuna, Itabuna, Estado de Bahia
  - Salvador, Salvador, Estado de Bahia
  - Teresina, Teresina, Piauí
  - Natal, Natal, Rio Grande do Norte
  - Ijuí, Ijuí, Rio Grande do Sul
  - Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Joinville, Joinville, Santa Catarina
  - São José Do Rio Preto, São José do Rio Preto, São Paulo
  - Curitiba, Curitiba
- Canada (8):
  - Calgary, Calgary, Alberta
  - Vancouver, Vancouver, British Columbia
  - Halifax, Halifax, Nova Scotia
  - Hamilton, Hamilton, Ontario
  - London, London, Ontario
  - Montreal, Montreal, Quebec
  - Sherbrooke, Sherbrooke, Quebec
  - Quebec, Québec
- China (12):
  - Nanjing, Nanjing, Jiangsu
  - Changchun, Changchun, Jilin
  - Shanghai, Shanghai, Shanghai Municipality
  - Taiyuan, Taiyuan, Shanxi
  - Beijing, Beijing
  - Beijing Shi, Beijing
  - Chongqing, Chongqing
  - Hangzhou, Hangzhou
  - Lanzhou, Lanzhou
  - Nanchang, Nanchang
  - Shanghai, Shanghai
  - Suzhou, Suzhou
- Denmark (4):
  - Alborg, Aalborg
  - Aarhus, Aarhus
  - Herlev, Herlev
  - Vejle, Vejle
- Finland (4):
  - Helsinki, Helsinki
  - Seinajoki, Seinäjoki
  - Tampere, Tampere
  - Turku, Turku
- France (4):
  - Strasbourg, Strasbourg, Bas-Rhin
  - Pierre Benite, Pierre-Bénite, Rhone
  - Creteil, Créteil, Val-de-Marne
  - Lyon, Lyon
- Germany (6):
  - Emmendingen, Emmendingen, Baden-Wurttemberg
  - Planegg, Planegg, Bavaria
  - Braunschweig, Braunschweig, Lower Saxony
  - Dresden, Dresden
  - Lubeck, Lübeck
  - Munster, Münster
- Italy (7):
  - Meldola, Meldola, Emilia-Romagna
  - Rome, Rome, Lazio
  - Cremona, Cremona, Lombardy
  - Candiolo, Candiolo, Piedmont
  - Orbassano, Orbassano, Piedmont
  - Arezzo, Arezzo, Tuscany
  - Milano, Milan
- Japan (19):
  - Kanazawa-shi, Kanazawa, Ishikawa-ken
  - Yokohama, Yokohama, Kanagawa
  - Sendai, Sendai, Miyagi
  - Osaka-sayama, Ōsaka-sayama, Osaka
  - Suita, Suita, Osaka
  - Bunkyō-Ku, Bunkyō-Ku, Tokyo
  - Nakano-ku, Nakano-ku, Tokyo
  - Sumida-ku, Sumida-ku, Tokyo
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Hiroshima, Hiroshima
  - Kita-gun, Kita-ku
  - Kyoto, Kyoto
  - Maebashi, Maebashi
  - Nagasaki, Nagasaki
  - Osaka, Osaka
  - Sapporo, Sapporo
  - Tokyo, Tokyo
  - Ube, Ube
- Netherlands (3):
  - Eindhoven, Eindhoven, North Brabant
  - Amsterdam, Amsterdam, North Holland
  - Sneek, Sneek
- New Zealand (4):
  - Christchurch, Christchurch
  - Dunedin, Dunedin
  - Hamilton, Hamilton
  - Tauranga, Tauranga
- Poland (5):
  - Lublin, Lublin, Lublin Voivodeship
  - Siedlce, Siedlce, Masovian Voivodeship
  - Warszawa, Warsaw, Masovian Voivodeship
  - Gdynia, Gdynia, Pomeranian Voivodeship
  - Katowice, Katowice
- Slovakia (8):
  - Bratislava, Bratislava
  - Kosice, Košice
  - Martin, Martin
  - Nitra, Nitra
  - Poprad, Poprad
  - Presov, Prešov
  - Sala, Šaľa
  - Trencin, Trenčín
- South Korea (5):
  - Goyang-Si, Goyang-si, Gyeonggido
  - Busan, Busan
  - Daegu, Daegu
  - Hwasun, Hwasun
  - Seoul, Seoul
- Spain (6):
  - A Coruna, A Coruña, A Coruna
  - Oviedo, Oviedo, Principality of Asturias
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Salamanca, Salamanca
  - Valencia, Valencia
- Sweden (4):
  - Orebro, Örebro, Orebro Ian
  - Stockholm, Stockholm, Sodermandlands Ian
  - Uppsala, Uppsala, Uppsala County
  - Malmo, Malmo
- Taiwan (2):
  - Kaohsiung City, Kaohsiung City
  - Taipei, Taipei
- United Kingdom (4):
  - Exeter, Exeter, Devon
  - Scunthorpe, Scunthorpe, North Lincolnshire
  - Nottingham, Nottingham
  - Rhyl, Rhyl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shore ND, Saad F, Cookson MS, George DJ, Saltzstein DR, Tutrone R, Akaza H, Bossi A, van Veenhuyzen DF, Selby B, Fan X, Kang V, Walling J, Tombal B; HERO Study Investigators. Oral Relugolix for Androgen-Deprivation Therapy in Advanced Prostate Cancer. N Engl J Med. 2020 Jun 4;382(23):2187-2196. doi: 10.1056/NEJMoa2004325. Epub 2020 May 29. PMID 32469183
- [Derived] Shore ND, Mehlhaff BA, Cookson MS, Saltzstein DR, Tutrone R, Brown B, Lu S, Fallick M, Hanson S, Saad F. Impact of Concomitant Cardiovascular Therapies on Efficacy and Safety of Relugolix vs Leuprolide: Subgroup Analysis from HERO Study in Advanced Prostate Cancer. Adv Ther. 2023 Nov;40(11):4919-4927. doi: 10.1007/s12325-023-02634-7. Epub 2023 Sep 15. PMID 37713020
- [Derived] Shore ND, Sutton J. Plain language summary of the HERO study comparing relugolix with leuprolide for men with advanced prostate cancer. Future Oncol. 2022 Jul;18(21):2575-2584. doi: 10.2217/fon-2022-0172. Epub 2022 May 19. PMID 35587650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To support registration in China, the study continued to enroll additional nonmetastatic or metastatic participants from China after the final analysis to reach the target enrollment of approximately 90 participants.
Pre-assignment Details: The primary analysis of efficacy and safety included 934 participants. The primary analysis excluded additional participants with metastatic disease and a cohort of participants enrolled in China and Taiwan who will be included in the final analysis of the study (N=200).
Groups:
- Relugolix: Relugolix 120-milligram (mg) tablet administered orally once daily for 48 weeks following an oral loading dose of 360 mg (3 x 120-mg tablets) on Day 1.
- Leuprolide Acetate: Leuprolide acetate depot suspension, 22.5 mg (or 11.25 mg in Japan and Taiwan), every 3 months by subcutaneous injection.
Period: Overall Study
Arm/Group | Relugolix | Leuprolide Acetate
Started | 624 | 310
Received at Least 1 Dose of Study Drug (Four participants (2 in each treatment group) were randomized but did not receive study drug.) | 622 | 308
Completed (Completed 48 weeks of treatment.) | 563 | 276
Not Completed | 61 | 34
Not completed — Adverse Event | 23 | 8
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 17 | 6
Not completed — Physician Decision | 9 | 3
Not completed — Testosterone Suppression Level Not Met | 7 | 13
Not completed — Did not Receive Study Drug | 2 | 2
Not completed — Dosing Interruption (Logistical Reason) | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug in the primary analysis part of the study.
Groups:
- Relugolix: Relugolix 120-mg tablet administered orally once daily for 48 weeks following an oral loading dose of 360 mg (3 x 120-mg tablets) on Day 1.
- Total: Total of all reporting groups
Arm/Group | Relugolix | Leuprolide Acetate | Total
Number analyzed (Participants) | 622 | 308 | 930
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (7.75) | 71.0 (8.03) | 71.1 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 622 | 308 | 930
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 31 | 83
  Not Hispanic or Latino | 558 | 269 | 827
  Unknown or Not Reported | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 127 | 71 | 198
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 16 | 46
  White | 434 | 202 | 636
  More than one race | 11 | 4 | 15
  Unknown or Not Reported | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Sustained Castration Rate
Description: Sustained castration rate defined as the cumulative probability of testosterone suppression to < 50 nanogram (ng)/deciliter (dL). The rate was estimated for each treatment group using the Kaplan-Meier method and reported as percentage of participants.
  The lower bound of the 95% confidence interval (CI) for the cumulative probability of sustained testosterone suppression in the relugolix treatment group must have been ≥ 90% to meet evaluation criteria for efficacy.
Time Frame: From Week 5 Day 1 (Day 29) to Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 96.7 [94.9 to 97.9] | 88.8 [84.6 to 91.8]
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Following statistical analysis of the lower bound of the 95% CI ≥ 90% for the relugolix group, secondary statistical analysis of non-inferiority was conducted; Test type: Non-Inferiority — The lower bound of the 95% CI for the difference in the cumulative probability of sustained profound castration rate between the 2 treatment groups was calculated with a noninferiority margin of -10%; Treatment difference = 7.9, 95% CI 2-sided [4.1 to 11.8] — Treatment difference= Relugolix - Leuprolide acetate
Statistical Analysis 2: Comparison: Relugolix vs Leuprolide Acetate; Following statistical analysis of the lower bound of the 95% CI ≥ 90% for the relugolix group, secondary statistical analysis of superiority was conducted; Test type: Superiority — If non-inferiority was demonstrated, superiority could be claimed if the lower bound of the 95% CI for the difference in the cumulative probability of sustained profound castration rate between the 2 treatment groups also excluded 0%. The p value was calculated post hoc; p < 0.0001, t-test, 2 sided; Two-sided type I error of 0.05

2. Secondary Outcome: Castration Rate At Week 1 Day 4
Description: Castration rate was defined as the cumulative probability of testosterone suppression to < 50 ng/dL. The rate was estimated for each treatment group using the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Week 1 Day 4 (Day 4)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 56.04 [52.18 to 59.97] | 0.00 [NA to NA] — Not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Alpha-protected statistical analysis; Test type: Superiority; p < 0.0001, t-test, 2 sided — Statistically significance was met if p-value < 0.05; Two-sided type I error rate of 0.05

3. Secondary Outcome: Castration Rate At Week 3 Day 1
Description: as for outcome 2
Time Frame: Week 3 Day 1 (Day 15)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 98.71 [97.56 to 99.39] | 12.05 [8.88 to 16.25]
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Alpha-protected statistical analysis; Test type: Superiority; p < 0.0001, t-test, 2 sided — Statistically significance was met if p-value < 0.05; Two-sided type I error rate of 0.05

4. Secondary Outcome: Confirmed Prostate-specific Antigen (PSA) Response Rate
Description: Confirmed PSA response defined as > 50% reduction in PSA from baseline at Week 3 Day 1 followed with confirmation at Week 5 Day 1.
Time Frame: Week 3 Day 1 (Day 15) and Week 5 Day 1 (Day 29)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 79.4 [76.03 to 82.53] | 19.8 [15.50 to 24.70]
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Alpha-protected statistical analysis; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Statistically significance was met if p-value < 0.05

5. Secondary Outcome: Profound Castration Rate At Week 3 Day 1 (Day 15)
Description: Castration rate defined as the cumulative probability of testosterone suppression to < 20 ng/dL. The rate was estimated for each treatment group using the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Week 3 Day 1 (Day 15)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 78.38 [75.06 to 81.53] | 0.98 [0.32 to 3.00]
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Alpha-protected statistical analysis; Test type: Superiority; p < 0.0001, t-test, 2 sided — Statistically significance was met if p-value < 0.05; Two-sided type I error rate of 0.05; Treatment difference = 77.41, 95% CI 2-sided [73.98 to 80.83] — Treatment difference= Relugolix - Leuprolide acetate

6. Secondary Outcome: Follicle-stimulating Hormone (FSH) Level
Description: To evaluate the effect of relugolix and leuprolide acetate on FSH suppression.
Time Frame: Week 25 Day 1 (Day 169)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
IU/L | 1.72 (1.376) | 5.95 (3.071)
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Alpha-protected statistical analysis; Test type: Superiority; p < 0.0001, t-test, 2 sided — Statistically significance was met if p-value < 0.05; Two-sided type I error rate of 0.05

7. Secondary Outcome: PSA Response Rate At Week 3 Day 1
Description: PSA response defined as > 50% reduction in PSA from baseline. The rate was estimated for each treatment group using the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Week 3 Day 1 (Day 15)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 80.1 [76.70 to 83.14] | 20.1 [15.80 to 25.05]

8. Secondary Outcome: PSA Response Rate At Week 5 Day 1
Description: as for outcome 7
Time Frame: Week 5 Day 1 (Day 29)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 94.5 [92.44 to 96.19] | 79.2 [74.26 to 83.61]

9. Secondary Outcome: Testosterone Recovery Rate
Description: The cumulative probability of testosterone recovery back to > 280 ng/dL (lower limit of the normal range), back to ≥ 50 ng/dL (definition of castration), and back to > 280 ng/dL or baseline at 90 days after drug discontinuation was assessed. The rate was estimated for each treatment group using the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Day 90 follow-up
Population: All randomized participants who received at least 1 dose of study drug and were followed in the testosterone recovery phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants
  ≥ 50 ng/dL | 93.01 [87.82 to 96.54] | 10.12 [3.84 to 25.24]
  > 280 ng/dL | 53.93 [45.20 to 63.16] | 3.23 [0.46 to 20.77]
  > Baseline level or 280 ng/dL | 54.73 [45.97 to 63.94] | 3.23 [0.46 to 20.77]

10. Secondary Outcome: Sustained Profound Castration Rate From Week 5 Day 1 Through Week 49 Day 1
Description: Sustained profound castration rate was defined as the cumulative probability of testosterone suppression to < 20 ng/dL. The rate was estimated by the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Week 5 Day 1 (Day 29) through Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 81.6 [78.1 to 84.5] | 68.6 [63.0 to 73.5]
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Test type: Other; Treatment difference = 13.0, 95% CI 2-sided [6.9 to 19.1] — Treatment difference= Relugolix - Leuprolide acetate

11. Secondary Outcome: Profound Castration Rate At Week 1 Day 4 (Day 4)
Description: as for outcome 5
Time Frame: At Week 1 Day 4 (Day 4)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 6.92 [5.18 to 9.22] | 0.0 [NA to NA] — Not estimable due to insufficient number of participants with events.

12. Secondary Outcome: Sustained Profound Castration Rate From Week 25 Day 1 Through Week 49 Day 1
Description: as for outcome 10
Time Frame: Week 25 Day 1 (Day 169) through Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug and had analyzable data at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 84.6 [81.3 to 87.3] | 87.5 [83.0 to 90.8]
Statistical Analysis 1: Comparison: Relugolix vs Leuprolide Acetate; Test type: Other; Treatment difference = -2.9, 95% CI 2-sided [-7.8 to 2.0] — Treatment difference= Relugolix - Leuprolide acetate

13. Secondary Outcome: Undetectable PSA Rate
Description: Defined as the proportion of participants with PSA concentration < 0.02 ng/milliliter (mL).The rate was estimated by the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Week 25 Day 1 (Day 169)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 20.7 [17.62 to 24.14] | 20.8 [16.39 to 25.74]

14. Secondary Outcome: Rate Of PSA Progression-free Survival
Description: PSA progression was defined as the first increase in PSA of 25% or greater and 2 ng/mL or greater above the nadir with confirmation by a second consecutive PSA measurement at least 3 weeks later. For participants without declining PSA from baseline, a PSA increase of ≥ 25% and ≥ 2 ng/mL from baseline beyond 12 weeks was considered PSA progression. The rate of progression-free survival was estimated using the Kaplan-Meier method and reported as percentage of participants.
Time Frame: Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 89.31 [86.52 to 91.55] | 89.50 [85.39 to 92.50]

15. Secondary Outcome: Change From Baseline In Quality Of Life (QoL) Total Score As Assessed By The Global Health Domain Of The European Organisation Of Research And Treatment Of Cancer (EORTC)-Quality Of Life Questionnaire (QLQ)-C30
Description: The EORTC QLQ-C30 core measurement was used to capture distal outcomes, including physical, social functioning, and overall health-related quality of life. The questionnaire incorporates 30 questions comprising nine multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 3 symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality of life scale. All raw domain scores are linearly transformed to a 0-100 scale. The global health and quality of life domain is presented. An increase in activity or functioning scores indicates improvement (higher/healthier level of functioning) and a decrease in symptom scores indicates improvement (lower level of symptoms/problems).
Time Frame: Baseline, Week 49 Day 1 (Day 337)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 543 | 257
score on a scale | -3.8 (18.13) | -3.6 (15.70)

16. Secondary Outcome: Change From Baseline In QoL Total Score For Remaining Domain Scores As Assessed By The EORTC-QLQ-C30
Description: The EORTC QLQ-C30 core measurement was used to capture distal outcomes, including physical, social functioning, and overall health-related quality of life. The questionnaire incorporates 30 questions comprising nine multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 3 symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality of life scale. All raw domain scores are linearly transformed to a 0-100 scale. All domains except for the global health and quality are presented. An increase in activity or functioning scores indicates improvement (higher/healthier level of functioning) and a decrease in symptom scores indicates improvement (lower level of symptoms/problems).
Time Frame: Baseline, Week 49 Day 1 (Day 337)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 543 | 257
score on a scale
  Physical functioning | -4.6 (13.09) | -4.4 (12.29)
  Role functioning | -6.2 (19.92) | -5.6 (17.84)
  Emotional functioning | 0.5 (16.12) | -0.5 (13.23)
  Cognitive functioning | -3.7 (16.77) | -3.8 (16.37)
  Social functioning | -2.7 (18.31) | -4.0 (18.18)
  Fatigue | 6.1 (19.46) | 7.0 (18.40)
  Nausea and vomiting | 0.2 (7.12) | 0.8 (6.02)
  Pain | 1.7 (20.19) | 4.0 (21.96)
  Dyspnoea | 5.3 (19.16) | 7.9 (20.25)
  Insomnia | 4.8 (25.88) | 4.8 (21.82)
  Appetite loss | -0.6 (17.82) | -0.6 (14.86)
  Constipation | 1.4 (23.26) | 3.5 (18.88)
  Diarrhoea | 2.0 (16.70) | 1.4 (19.60)
  Financial difficulties | 0.2 (18.28) | 0.1 (19.21)

17. Secondary Outcome: Change From Baseline In QoL Total Score As Assessed By The EORTC-QLQ-PR25 Sexual Activity And Functioning And Hormonal-Treatment-Related Symptom Subdomains
Description: Subscales for assessment of hormonal treatment-related symptoms (6 items) and sexual activity and function (6 items) from the EORTC-QLQ-PR25 25-item prostate cancer module of the EORTC are presented. Questions used 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale. An increase in activity or functioning scores indicates improvement (higher/healthier level of functioning) and a decrease in symptom scores indicates improvement (lower level of symptoms/problems).
Time Frame: Baseline, Week 49 Day 1 (Day 337)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 537 | 256
score on a scale
  Sexual activity | 13.9 (26.51) | 10.8 (27.90)
  Sexual functioning | -9.0 (23.37) | -10.4 (21.10)
  Hormonal treatment-related symptoms | 10.6 (12.25) | 11.4 (13.30)

18. Secondary Outcome: Change From Baseline In QoL Total Score For Urinary And Bowel Symptoms Domains As Assessed By The EORTC-QLQ-PR25
Description: Subscale assessments of urinary symptoms (9 items) and bowel symptoms (4 items) from the EORTC-QLQ-PR25 25-item prostate cancer module of the EORTC are presented. Questions used 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale. A decrease in symptom scores indicates improvement (lower level of symptoms/problems).
Time Frame: Baseline, Week 49 Day 1 (Day 337)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 537 | 256
score on a scale
  Urinary symptoms | 1.1 (15.29) | -0.4 (13.78)
  Incontinence aid use | 1.0 (15.41) | 0.0 (19.80)
  Bowel symptoms | 1.2 (8.92) | 2.0 (9.51)

19. Secondary Outcome: Change From Baseline In QoL Total Score As Assessed By The European Quality Of Life 5-Dimension 5-Level Questionnaire (EuroQoL EQ-5D-5L)
Description: The EuroQoL EQ-5D-5L comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 levels: no problems (1 as numerical score), slight problems (2 as numerical score), moderate problems (3 as numerical score), severe problems (4 as numerical score), and extreme problems (5 as numerical score). The total score ranges from 0 to 100. A decrease in score indicates improvement.
Time Frame: Baseline, Week 49 Day 1 (Day 337)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 549 | 259
score on a scale | -1.5 (14.36) | -2.7 (14.57)

20. Secondary Outcome: Percent Change From Baseline In Serum Concentrations Of Luteinizing Hormone
Description: Blood samples were collected from participants for hormonal measurements.
Time Frame: Week 1 Day 4 (Day 4), Week 5 Day 1 (Day 29), Week 25 Day 1 (Day 169), and Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
Percent change
  Week 1 Day 4 (Day 4) | -88.25 (20.696) | 147.71 (122.735)
  Week 5 Day 1 (Day 29) | -94.54 (8.500) | -82.67 (27.146)
  Week 25 Day 1 (Day 169) | -93.93 (7.242) | -93.45 (13.202)
  Week 49 Day 1 (Day 337) | -91.54 (16.779) | -95.14 (4.507)

21. Secondary Outcome: Percent Change From Baseline In Serum Concentrations Of FSH
Description: Blood samples were collected from participants for hormonal measurements.
Time Frame: Week 1 Day 4 (Day 4), Week 5 Day 1 (Day 29), Week 25 Day 1 (Day 169), and Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percent change
  Week 1 Day 4 (Day 4) | -62.59 (9.051) | -4.74 (36.121)
  Week 5 Day 1 (Day 29) | -90.80 (8.151) | -67.73 (27.311)
  Week 25 Day 1 (Day 169) | -86.32 (10.699) | -47.53 (32.560)
  Week 49 Day 1 (Day 337) | -79.39 (21.987) | -47.23 (30.112)

22. Secondary Outcome: Percent Change From Baseline In Serum Concentrations Of Dihydrotestosterone
Description: Blood samples were collected from participants for hormonal measurements.
Time Frame: Week 5 Day 1 (Day 29), Week 25 Day 1 (Day 169), and Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percent change
  Week 5 Day 1 (Day 29) | -87.61 (12.225) | -81.95 (23.733)
  Week 25 Day 1 (Day 169) | -88.06 (11.810) | -85.45 (32.261)
  Week 49 Day 1 (Day 337) | -88.23 (11.235) | -87.56 (12.088)

23. Secondary Outcome: Percent Change From Baseline In Serum Concentrations Of Sex Hormone-Binding Globulin
Description: Blood samples were collected from participants for hormonal measurements.
Time Frame: Week 5 Day 1 (Day 29), Week 25 Day 1 (Day 169), and Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percent change
  Week 5 Day 1 (Day 29) | 1.08 (22.068) | -1.21 (20.430)
  Week 25 Day 1 (Day 169) | 7.24 (28.265) | 3.59 (24.947)
  Week 49 Day 1 (Day 337) | 6.54 (28.787) | 2.59 (27.051)

24. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Of Relugolix
Description: The Cmax of relugolix was determined for single and repeat doses in subsets of participants from Japan. Single dose pharmacokinetics (PK) was assessed on Day 1 following an initial 360 mg dose of relugolix. Repeat dose PK was assessed following repeat dosing of relugolix 120 mg once daily for 2 weeks.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hours postdose on Day 1 and Week 2
Population: A subset of Japanese participants enrolled in study were included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Relugolix Single-Dose: Relugolix oral loading dose of 360 mg (3 x 120-mg tablets) on Day 1.
- Relugolix Repeat-Dose: Relugolix 120-mg tablet administered orally once daily for 2 weeks following an oral loading dose of 360 mg (3 x 120-mg tablets) on Day 1.
Arm/Group | Relugolix Single-Dose | Relugolix Repeat-Dose
Number analyzed (Participants) | 7 | 7
ng/mL | 125 (220) | 46.4 (141)

25. Secondary Outcome: Area Under The Concentration-Time Curve (AUC0-τ) Of Relugolix
Description: The AUC0-τ of relugolix was determined for single and repeat doses in subsets of participants from Japan. Single dose PK was assessed on Day 1 following an initial 360 mg dose of relugolix. Repeat dose PK was assessed following repeat dosing of relugolix 120 mg once daily for 2 weeks.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hours postdose on Day 1 and Week 2
Population: A subset of Japanese participants enrolled in study were included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng⸳hr/mL
Arm/Group | Relugolix Single-Dose | Relugolix Repeat-Dose
Number analyzed (Participants) | 7 | 7
ng⸳hr/mL | 663 (151) | 373 (51)

26. Secondary Outcome: Time To Maximum Observed Plasma Concentration (Tmax) Of Relugolix
Description: The Tmax of relugolix was determined for single and repeat doses in subsets of participants from Japan. Single dose PK was assessed on Day 1 following an initial 360 mg dose of relugolix. Repeat dose PK was assessed following repeat dosing of relugolix 120 mg once daily for 2 weeks.
Time Frame: Predose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hours postdose on Day 1 and Week 2
Population: A subset of Japanese participants enrolled in study were included in the PK analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Relugolix Single-Dose | Relugolix Repeat-Dose
Number analyzed (Participants) | 7 | 7
hours | 1.03 [0.400 to 4.05] | 0.983 [0.433 to 4.08]

27. Other Pre Specified Outcome: Percentage of Participants Who Experienced Major Adverse Cardiovascular Events (MACE)
Description: MACE were defined as nonfatal myocardial infarction, nonfatal stroke, and death from any cause.
Time Frame: From Week 5 Day 1 (Day 29) to Week 49 Day 1 (Day 337)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix | Leuprolide Acetate
Number analyzed (Participants) | 622 | 308
percentage of participants | 2.9 | 6.2

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through up to 52 weeks
Description: All randomized participants who received at least 1 dose of study drug in the primary analysis part of the study.
Groups:
- Leuprolide Acetate: Leuprolide acetate depot suspension, 22.5 mg (or 11.25 mg in Japan, and Taiwan), every 3 months by subcutaneous injection.
Arm/Group | Relugolix | Leuprolide Acetate
All-Cause Mortality (participants affected / at risk) | 7/622 | 9/308
Serious Adverse Events (participants affected / at risk) | 76/622 | 47/308
Other Adverse Events (participants affected / at risk) | 493/622 | 239/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix (N=622) | Leuprolide Acetate (N=308)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 3
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Appendicitis perforated (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Shunt aneurysm (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Mental disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Bladder obstruction (Renal and urinary disorders) | 2 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Homicide (Social circumstances) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix (N=622) | Leuprolide Acetate (N=308)
Constipation (Gastrointestinal disorders) | 76 | 30
Diarrhoea (Gastrointestinal disorders) | 76 | 21
Nausea (Gastrointestinal disorders) | 36 | 13
Asthenia (General disorders) | 32 | 21
Fatigue (General disorders) | 134 | 57
Nasopharyngitis (Infections and infestations) | 59 | 29
Weight increased (Investigations) | 49 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 | 19
Dizziness (Nervous system disorders) | 35 | 17
Headache (Nervous system disorders) | 35 | 13
Insomnia (Psychiatric disorders) | 43 | 14
Nocturia (Renal and urinary disorders) | 36 | 19
Pollakiuria (Renal and urinary disorders) | 37 | 20
Urinary incontinence (Renal and urinary disorders) | 30 | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 | 16
Hot flush (Vascular disorders) | 338 | 159
Hypertension (Vascular disorders) | 49 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03085095/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03085095/SAP_000.pdf